CLINICAL TRIAL: NCT06478381
Title: A Phase 1, Open-label, Dose Escalating Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of L218CAR19 in Patients With CD19 Positive Relapsed/Refractory B-cell Lymphomas
Brief Title: L218CAR19 in Patients With Relapsed/Refractory B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanyan Liu, Professor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYML09
Record Dates: First submitted 2024-06-16; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Relapsed/Refractory B-cell Lymphomas
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): L218CAR19 is administered via infusion with ascending dose levels to determine the maximum tolerated dose (MTD)
  Interventions: Drug: L218CAR19

INTERVENTIONS:
Drug: L218CAR19 — L218CAR19 is intravenously administered at three dose levels.

SUMMARY:
L218CAR19 is a kind of chimeric antigen receptor T-cell immunotherapy targeting CD19 on B cells. The goal of this study is to determine the safety, tolerability, pharmacokinetics, pharmacodynamics and clinical activity of L218CAR19 in patients with B-cell lymphomas who have received at least two lines of systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years at the time of inclusion
* Written informed consent
* Patients with relapsed/refractory CD19 positive B-cell lymphomas, who have received at least two lines of treatment
* With measurable disease
* ECOG PS 0-2 at protocol entry
* Estimated life expectancy of 3 months or longer
* Hemoglobin ≥ 8 g/dL (≥5 mmol/l); Platelets ≥ 75 x 10E9/L; Absolute neutrophil count ≥ 1.0 x 10E9/L; Platelets ≥ 50 x 10E9/L permitted if documented bone marrow involvement; Serum bilirubin ≤ 1.5 x upper limit of normal (ULN), or ≤3 x ULN if elevation is due to hepatic involvement by lymphoma; Serum glutamic-oxaloacetic transaminase (AST) and/or serum glutamic-pyruvic transaminase (ALT) ≤ 2.5 x ULN, or ≤ 5 x ULN if elevation is due to hepatic involvement by lymphoma; Serum creatinine ≤ 1.5 x ULNb; left ventricular ejection fraction (LVEF) ≥ 50%
* Women of childbearing potential must use safe anticonception (e.g. contraceptive pills, intrauterine devices etc.) during the study and 6 months after the administration of study drug; Male patients must use contraception for the duration of the study and 6 months after the administration of study drug if his partner is of childbearing potential

Exclusion Criteria:

* Patients with heart disease: atrial fibrillation; History of Class III or IV New York Heart Association (NYHA) heart failure, myocardial infarction or other significant cardiac disease within 12 months of screening; LVEF<50%; clinical significant pericardial effusion; Long QT syndrome
* History of severe pulmonary function impairment
* With other uncontrolled malignancy
* With active bacterial, viral, or fungal infections
* WIth uncontrolled autoimmune disease or congential immunodeficiency
* HIV antibody positive patients
* Known severe hypersensitivity to biological product
* Patients with known active central nervous system (CNS) disease, including lymphoma CNS involvement
* Patients with prior CAR-T therapy
* History of allogeneic stem cell transplantation
* History of autogeneic stem cell transplantation within 6 months of screening
* History of major surgery within 4 weeks of screening
* Patients receiving live (attenuated) vaccines within 6 weeks of screening
* Pregnant or lactating women, or pregnant plan within 12 months
* Involvement of cardiac tissue by lymphoma
* with emergency due to oncothlipsis
* Unwillingness or inability to comply with the protocol
* Deemed 'unfit' by the treating physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 4 weeks
  Occurrence of DLTs
Treatment-emergent adverse event (AE) | Up to 1 year
  Incidence of treatment-emergent AEs

SECONDARY OUTCOMES:
Quantification of L218CAR19 in peripheral blood | Up to 1 year
  To quantify L218CAR19 in a patient's peripheral blood at different time points
Time to reach Cmax (Tmax) of L218CAR19 | Up to 3 months
  To identify the time point when the concentration of L218CAR19 reaches maximum in a patient's peripheral blood
Area under the curve (AUC) of L218CAR19 | Up to 3 months
  To quantify the cumulative amount of L218CAR19 in a patient's peripheral blood over time
Clearance (CL) of L218CAR19 | Up to 3 months
  To determine the clearance factor of L218CAR19 in a patient's peripheral blood
Immunogenic response to L218CAR19 | Up to 1 year
  To evaluate the anti-drug antibodies in response to L218CAR19 administration in a patient's peripheral blood
Serum cytokine concentrations | Up to 3 months
  To measure the cytokine levels (e.g. TNFa, IL-6, IL-1, IL-2, etc.) in a patient's peripheral blood at different time points
ORR | Up to 1 year
  To determine the overall (best) objective anti-cancer response by Lugano criteria
PFS | Up to 1 year
  To evaluate the duration of patient's progression-free survival
OS | Up to 1 year
  To evaluate the overall duration of patient's survival

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, Principal Investigator — Affiliated Cancer Hospital of Zhengzhou University
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan, China